CLINICAL TRIAL: NCT06297863
Title: Head Down Tilt 15° to Increase Collateral Flow in Acute Ischemic Stroke: a Multicenter, Randomised, Proof of Concept, Phase 2a/b Trial in Patients Treated With Mechanical Thrombectomy
Brief Title: Head Down Tilt 15° to Increase Collateral Flow in Acute Ischemic Stroke
Acronym: DOWN-SUITE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Fondazione IRCCS San Gerardo dei Tintori (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other); Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other); Università degli Studi dell'Aquila (Other); Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOWN-SUITE
Record Dates: First submitted 2024-02-26; First posted 2024-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
Keywords: Collaterals; Cerebral hemodynamics; Head down positioning
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: The DOWN-SUITE trial is a prospective, multicenter, proof of concept, randomised, controlled, open label, phase 2a/b clinical trial with blinded outcome assessment, comparing cerebral collateral status in patients with acute ischemic stroke due to middle cerebral artery occlusion (M1 segment) treated with in-hospital application of HDT15 (-10° to -15°) versus usual positioning (0° to +30°), before and during mechanical thrombectomy.
Who Masked: Outcomes Assessor
Masking Description: A blinded central imaging core lab, whose members will be unaware of the procedure assignments, will assess all imaging outcomes, including the primary efficacy outcome (collateral status, assessed during the pretreatment diagnostic angiographic series of mechanical thrombectomy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEAD DOWN TILT -10° to -15° (HDT15) (Experimental): HDT15 will be applied in the intervention group in 2 different settings:
  * in the Emergency Room, by tilting the stretcher to lower the head by -10° to -15° relative to the body of the patient; the degree of tilting will be checked using a dedicated digital inclinometer or a mobile phone app
  * in the Angiography Suite, by tilting the angiography table to lower the head by -10° to -15° relative to the body of the patient, depending on the actual technology of the angiography system of each clinical site; the degree of tilting will be automatically checked using the angiography system HDT15 will start as soon as possible following randomisation in the Emergency Room (i.e. after vascular neuroimaging), and will be maintained during the transfer to the Angiography Suite, as well as during the entire thrombectomy procedure. HDT15 will end after the completion of mechanical thrombectomy.
  Interventions: Procedure: HEAD DOWN TILT -10° to -15°
- USUAL POSITIONING (No Intervention): Patients randomised in the control group will be maintained in the usual position during the emergency room phase (0° to +30°) and on the angiography table (0°), according to standard practice. Mechanical thrombectomy will be performed as per usual care.

INTERVENTIONS:
Procedure: HEAD DOWN TILT -10° to -15° — Head down tilt -10° to -15° (HDT15) is a positional therapy consisting of tilting the patient with the head -10° to -15° degrees below the rest of the body.
  Application of HDT15 will not delay usual care. The standard in-hospital patient pathway, including transfer from neuroimaging room to the angiography suite and the required procedural steps of MT, will allow sufficient time for the application of HDT15. HDT15 duration is expected to be at least 30 minutes (estimated time 30 to 90 minutes), from start to the assessment of the primary efficacy endpoint.
  The actual degree of HDT15 will be a range between -10° to -15°, depending on the angiographic system of each clinical site, but it will be maintained at -15° during the Emergency Room phase which is expected to account for >50% of the total application time.
  Arms: HEAD DOWN TILT -10° to -15° (HDT15)

SUMMARY:
The DOWN-SUITE study is multicenter, randomised, controlled, open-label clinical trial with blinded outcome assessment comparing collateral status in patients with acute ischemic stroke treated with an in-hospital application of head down tilt -10° to -15° (HDT15) versus usual positioning (0° to +30°) before endovascular mechanical thrombectomy.

This study will involve adult patients who are eligible for mechanical thrombectomy and who have acute ischemic stroke due to left or right middle cerebral artery occlusion (M1 segment).

The investigators hypothesise that HDT15, applied in acute ischemic stroke patients with a large vessel occlusion, will improve collateral circulation, prolong the survival of the ischemic penumbra and improve the clinical benefit from mechanical thrombectomy compared with standard of care (usual positioning 0° to +30°).

DETAILED DESCRIPTION:
Investigating, developing and implementing a collateral therapeutic is a major objective in stroke research. The aim is to increase the amount of potentially salvageable penumbral tissue and expand the tissue time window, thus increasing the efficacy of reperfusion therapies and improving clinical outcomes.

Head down tilt 15° (HDT15) is a positional therapy consisting of tilting the patient with the head 15 degrees below the rest of the body. Experimental studies from an Italian-French group (Dr. Simone Beretta, Fondazione IRCCS San Gerardo dei Tintori and Prof. Tae-Hee Cho, Hospices Civils de Lyon) showed that HDT15 increased cerebral blood flow and improved functional outcome and infarct volume in randomised rats with middle cerebral artery (MCA) occlusion followed by reperfusion. Subsequent perfusion MRI experiments using the same stroke model by our group confirmed that HDT15 application for 60 minutes significantly increases collateral flow in the ischemic area.

There is no consensus in current clinical practice regarding the most appropriate head position for acute ischemic stroke (AIS) patients. The sitting position at +30° is the most common. An international cluster-randomised trial, HeadPoST, randomised over 11000 patients with acute stroke (85% ischemic) to either a lying-flat position or a sitting-up position (head elevated to at least 30°), maintained for 24 hours. No difference in the primary efficacy outcome (disability at 90 days measured with the modified Rankin Scale (mRS)), mortality, or rates of other serious adverse events, including pneumonia, were observed. However, the HeadPoST trial primarily targeted patients with mild symptoms without a large vessel occlusion (LVO), who were randomised beyond the usual time window of reperfusion therapies.

One retrospective study (pre-thrombectomy era) compared two cohorts of AIS patients with a LVO: patients with a standard position (0 to 30°; N=119), versus those with a HDT15 position (0 to -15°; N=90). The results suggested that HDT15 promotes neurological improvement compared to the standard position. No difference in serious adverse events was observed between the two cohorts.

A recent randomized, pilot clinical trial showed promising results of -20° head down positioning on long-term disability and an excellent safety profile.

Thus, the available clinical evidence raised no safety concern for HDT15 in AIS patients, but data on its efficacy, notably among AIS patients treated by MT, remains insufficient. HDT15, for its simplicity, low cost and feasibility, might be an optimal collateral therapeutic candidate to prolong the survival of the ischemic penumbra and improve the clinical benefit from reperfusion therapies with disability reduction. HDT15 is readily feasible by Emergency Services in the prehospital phase of AIS, before reperfusion therapies.

The DOWN-SUITE study will be the first multicenter, randomised, controlled, open-label clinical trial with blinded outcome assessment comparing collateral status in patients with AIS treated with an in-hospital application of HDT15 versus usual positioning before MT. The duration of HDT15 application (approximately 60-90 minutes) is expected to be long enough to detect significant changes in cerebral hemodynamics. Building from preclinical experiments on rodent and non-human primate stroke models carried out by our French-Italian group, it will provide for the first time the translation of HDT15 efficacy on cerebral hemodynamics and clinical outcome from animal models to AIS patients.

No therapeutic intervention is currently available to enhance collaterals in AIS.

The DOWN-SUITE trial will provide robust, high-quality evidence on the safety, feasibility and efficacy of HDT15 as a low-cost collateral therapeutic for AIS.

The investigators hypothesise that HDT15 (-10° to -15°), applied in AIS patients with an LVO, will improve collateral circulation, prolong the survival of the ischemic penumbra and improve the clinical benefit from MT compared with standard of care (usual positioning: 0° to +30°).

The investigators aim to perform a prospective, multicenter, proof of concept, randomised, controlled, open-label study. As a double-blind is not possible, a blinded central imaging core lab, whose members will be unaware of the procedure assignments, will assess all imaging outcomes, including the primary efficacy outcome.

This study will involve adult patients who are eligible for MT and who have AIS due to left or right MCA occlusion (M1 segment).

Benefit/risk ratio The investigators hypothesise that HDT15 would improve cerebral collaterals in patients randomised in the intervention group, which could subsequently reduce the ischemic injury and improve the clinical outcome.

No harm from participating in DOWN-SUITE is expected for patients in the intervention or control groups. Previous clinical data on HDT15 raised no safety concerns. No difference in post-stroke complications, including cerebral oedema or haemorrhage, pneumonia or mortality, was observed in a retrospective observational study. HDT15 is not expected to interfere with standard care, including the procedural steps of MT. Mild discomfort related to the tilted position may occur in some patients. The treating physician will continuously monitor all patients during the entire duration of the HDT15 application. No additional risk is expected in patients in the control group, as they will receive standard care.

Overall, this study's benefit/risk ratio is considered very favourable.

This study could potentially establish HDT15 as the first evidence-based collateral therapeutic for AIS. No therapeutic intervention is currently available to enhance collaterals in the acute phase of ischemic stroke. Such a collateral-enhancing therapy is necessary to expand the time window and increase the probability of successful reperfusion with IVT and MT, resulting in better clinical outcomes.

The results of the DOWN-SUITE trial may pave the way for larger randomised controlled trials of HDT15 in a wider stroke patient population, such as patients transferred from spoke hospitals to hub stroke centers to receive thrombectomy and unselected patients with suspected AIS in the prehospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke due to left or right MCA occlusion of the M1 segment (excluding occlusion of the internal carotid artery terminus + M1)
* Decision to treat with mechanical thrombectomy (with or without intravenous thrombolysis)
* Informed consent obtained from patient or patient's next of kin, or emergency consent procedure

Exclusion Criteria:

* Impaired consciousness, defined as NIHSS score of 2 or 3 of the item 1a (level of consciousness): not alert, requires repeated stimulation or unresponsive.
* Vomiting upon stroke onset.
* History of glaucoma.
* History or imaging findings of intracranial hypertension of any aetiology
* Major breath disorders, defined as follows:

  * oxygen saturation ≤92% in room air at admission
  * severe chronic obstructive pulmonary disease (COPD) treated with long-term oxygen therapy.
  * severe heart failure with NYHA class 3 or 4 (breathlessness during ordinary physical activity or at rest).
* Severe obesity, defined as body mass index (BMI) > 35.
* Patients participating in another interventional trial that would interfere with this study.
* Female patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Good collateral status | Day 0 (during mechanical thrombectomy)
  The primary endpoint will be the achievement of good collateral status, i.e. grade 3 or 4 on the American Society of Interventional and Therapeutic Neuroradiology/Society of Interventional Radiology (ASITN/SIR) collateral scale, in the HDT15 versus control group, as seen at the beginning of MT.15 The ASITN/SIR collateral grade will be assessed by a blinded central imaging core lab from the pretreatment diagnostic angiographic runs, routinely performed as the first procedural step of MT.

SECONDARY OUTCOMES:
Feasibility of HDT15 | Day 0 (in the emergency room and angio suite)
  proportion of patients randomised to the intervention group who are able to maintain HDT15 during the entire MT procedure
Delay to thrombectomy | Day 0 (in the emergency room and angio suite)
  hospital admission-to-arterial access time (i.e. time to arterial puncture)
Vomiting | Day 0 (in the emergency room and angio suite)
  Proportion of patients presenting one or more episodes of vomiting from randomisation to the completion of MT
Early neurological deterioration | 1 day (24±12 hours)
  Proportion of patients who had increase of ≥4 points on the NIHSS score within 24±12 hours of the randomisation
Symptomatic intracranial hemorrhage | 1 day (24±12 hours)
  Proportion of patients who had SICH per SITS-MOST definition within 24±12 hours: type 2 parenchymal hematoma with neurological deterioration of ≥4 points on the NIHSS
Aspiration pneumonia | 1 day (24±12 hours)
  Proportion of patients with pneumonia within the first 72 hours after randomisation
Neurological disability | 3 months
  functional outcome at 3 months, assessed with the ordinal score on the modified Rankin scale (shift across outcomes on the mRS between groups)
Systolic blood pressure | Day 0 (in the emergency room and angio suite)
  Mean values of systolic blood pressure (mmHg) from hospital admission to the end of MT; monitored at entry in the Emergency Room, at entry in the angio suite and every 15 minutes from the start to the end of MT
Diastolic blood pressure | Day 0 (in the emergency room and angio suite)
  Mean values of diastolic blood pressure (mmHg) from hospital admission to the end of MT; monitored at entry in the Emergency Room, at entry in the angio suite and every 15 minutes from the start to the end of MT
Oxygen saturation | Day 0 (in the emergency room and angio suite)
  Mean values of oxygen saturation (%) from hospital admission to the end of MT; these physiological parameters will be monitored at entry in the Emergency Room, at entry in the angio suite and every 15 minutes from the start to the end of MT

CONTACTS AND LOCATIONS:
Overall Officials: Simone Beretta, MD, PhD, Principal Investigator — University of Milano Bicocca
Locations (6):
- Italy (6):
  - Ospedale Civile SS. Nicola e Filippo Avezzano Pronto Soccorso, Avezzano
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera Policlinico Universitario "G. Martino", Messina
  - Fondazione IRCCS San Gerardo dei Tintori Monza, Monza
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
  - Ospedale Santa Maria della Misericordia, Udine

IPD SHARING:
Plan to Share IPD: Yes
The project data can be accessed by interested European and extra-EU third parties for replication or further analysis only if given in a completely anonymous form.
  Third parties in this project include academic institutions, research centers and non-profit associations (e.g. research consortia). Third parties in this project do not include profit associations (e.g. drug companies).
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After completion of the primary analysis
Access Criteria: If the need arises to communicate data in pseudo-anonymous form, the patient will, first of all, be informed and specific informed consent will be provided. In the latter case, the data will not be sent without the patient's consent. Ad hoc Data Transfer Agreements will be established with the interested third parties.

REFERENCES:
- [Background] Beretta S, Versace A, Carone D, Riva M, Dell'Era V, Cuccione E, Cai R, Monza L, Pirovano S, Padovano G, Stiro F, Presotto L, Paterno G, Rossi E, Giussani C, Sganzerla EP, Ferrarese C. Cerebral collateral therapeutics in acute ischemic stroke: A randomized preclinical trial of four modulation strategies. J Cereb Blood Flow Metab. 2017 Oct;37(10):3344-3354. doi: 10.1177/0271678X16688705. Epub 2017 Jan 23. PMID 28112023
- [Background] Diamanti S, Mariani J, Versace A, Riva M, Cuccione E, Cai R, Monza L, Vigano M, Bolbos R, Chauveau F, Cho TH, Carone D, Ferrarese C, Beretta S. Head down tilt 15 degrees to preserve salvageable brain tissue in acute ischemic stroke: A pre-clinical pooled analysis, with focus on cerebral hemodynamics. Eur J Neurosci. 2023 Jun;57(12):2149-2159. doi: 10.1111/ejn.15852. Epub 2022 Nov 4. PMID 36300727
- [Background] Anderson CS, Arima H, Lavados P, Billot L, Hackett ML, Olavarria VV, Munoz Venturelli P, Brunser A, Peng B, Cui L, Song L, Rogers K, Middleton S, Lim JY, Forshaw D, Lightbody CE, Woodward M, Pontes-Neto O, De Silva HA, Lin RT, Lee TH, Pandian JD, Mead GE, Robinson T, Watkins C; HeadPoST Investigators and Coordinators. Cluster-Randomized, Crossover Trial of Head Positioning in Acute Stroke. N Engl J Med. 2017 Jun 22;376(25):2437-2447. doi: 10.1056/NEJMoa1615715. PMID 28636854
- [Background] Gauthier A, Gerardin P, Renou P, Sagnier S, Debruxelles S, Poli M, Rouanet F, Olindo S, Sibon I. Trendelenburg Positioning in Large Vessel Ischaemic Stroke: A Pre-Post Observational Study Using Propensity Score Matching. Cerebrovasc Dis. 2018;46(1-2):24-32. doi: 10.1159/000490423. Epub 2018 Jul 27. PMID 30056454
- [Background] Chen HS, Zhang NN, Cui Y, Li XQ, Zhou CS, Ma YT, Zhang H, Jiang CH, Li RH, Wan LS, Jiao Z, Xiao HB, Li Z, Yan TG, Wang DL, Nguyen TN. A randomized trial of Trendelenburg position for acute moderate ischemic stroke. Nat Commun. 2023 May 5;14(1):2592. doi: 10.1038/s41467-023-38313-y. PMID 37147320